CLINICAL TRIAL: NCT06970860
Title: Detection of Bleeding Disorders Diagnosed After Vaginal Delivery Complicated by Severe Postpartum Hemorrhage
Acronym: DIDAPPH
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0169
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Severe Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; bleeding disorders
MeSH Terms: conditions — Postpartum Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The plasma bank will allow the measurement of biomarkers of interest.
  The DNA bank will also be used to validate the genetic polymorphisms that have been identified in association with severe PPH in another study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of women who experienced severe postpartum hemorrhage following a vaginal delivery.

SUMMARY:
A cohort study designed to detect bleeding disorders diagnosed in women who experienced severe postpartum hemorrhage after vaginal delivery

DETAILED DESCRIPTION:
Severe postpartum hemorrhage (PPH), defined as blood loss ≥ 1000 mL within 24 hours after delivery, is a common complication of childbirth (2% of deliveries in France and Europe). It is associated with significant maternal morbidity and mortality. Moreover, the incidence of PPH has been increasing in high-resource countries since the 1990s, making it a major public health issue.

Research conducted by our group on the Finistère cohort of pregnant women, highlighted that a first-degree family history of PPH is a risk factor for severe PPH after vaginal delivery, with an Odds Ratio of 2.37 (95% CI 1.56-3.60). These findings suggest a familial predisposition to PPH.

Furthermore, von Willebrand disease is the most common hereditary bleeding disorder worldwide, with an estimated prevalence between 0.6% and 1.3%. The most common form, type 1 von Willebrand disease, is inherited in an autosomal dominant manner.

There is limited data in the literature regarding the prevalence of bleeding disorders diagnosed following PPH in the general population. However, PPH is a frequent complication of childbirth in women with von Willebrand disease, with the prevalence of primary severe PPH being 2 to 4 times higher compared to the general population.

The research hypothesis of the DIDAPPH study is that severe PPH could be a presenting feature of previously undiagnosed von Willebrand disease.

If constitutional bleeding disorders were frequently diagnosed after severe PPH, then their systematic screening could be a public health priority for women of childbearing age and might enable more effective prevention of hemorrhagic complications during delivery, through prophylactic drug treatments, in subsequent pregnancies. Additionally, diagnosing von Willebrand disease in these women would have the added benefit of better preventing hemorrhagic complications after invasive procedures outside of pregnancy, particularly surgical ones, throughout their lifetime.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old
* Who experienced severe postpartum hemorrhage, defined as blood loss ≥ 1000 mL, following a vaginal delivery in the previous 12 months, in a maternity unit in Finistère

Exclusion Criteria:

* Women who are pregnant at the time of inclusion
* Women with a known hereditary bleeding disorder (Willebrand's disease, hemophilia carrier, etc.) or acute or chronic Immune thrombocytopenia (ITP) prior to delivery.
* Women with a known other bleeding pathology prior to delivery
* Women taking a treatment that interferes with hemostasis, such as aspirin, anticoagulants or non-steroidal anti-inflammatory drugs (biological sampling may be postponed until after the interfering treatment has stopped, in the case of occasional use of the latter).
* Women on long-term anticoagulant or antiaggregant therapy
* Women under legal protection,
* Women not affiliated to the French social security system.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The women included in the study will be adult women who experienced severe postpartum hemorrhage, defined as blood loss ≥1000 mL after a vaginal delivery. These women will be identified by the teams from the maternity units in Finistère.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2029-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of biological test results suggestive of a bleeding disorder, correlated with the clinical bleeding phenotype, within the cohort | From inclusion to three month

SECONDARY OUTCOMES:
Number of hereditary types of bleeding disorders diagnosed within the cohort based on the biological test results | From inclusion to three month
Number of acquired types of bleeding disorders within the cohort based on the biological test results | From inclusion to three month
Plasma levels of blood biomarkers associated with severe postpartum hemorrhage (PPH), as identified in another genetic study, among patients from the DIDAPPH cohort based on the biological test results | Inclusion
Frequency of genetic polymorphisms associated with severe postpartum hemorrhage identified in another genetic study among patients from the DIDAPPH cohort based on the biological test results | Inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.